CLINICAL TRIAL: NCT06541041
Title: Evaluation of Electrical Stimulation During Nerve Transfer Surgery for Cervical Spinal Cord Injury
Brief Title: Nerve Transfers Plus Electrical Stimulation to Improve Hand Function in Cervical Spinal Cord Injury
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas J Wilson, Clinical Professor, Stanford University
Other Study IDs: 75876
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Cervical Spinal Cord Injury; Cervical Spinal Cord Paralysis; Tetraplegia; Tetraplegia/Tetraparesis; Tetraplegic Spinal Paralysis
Keywords: Cervical Spinal Cord Injury; Nerve Transfer; Brief Intraoperative Electrical Stimulation; Peripheral Nerve Stimulation; Tetraplegia
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Arm A: Standard nerve transfer surgery without electrical stimulation: This is a retrospective group that has already undergone standard nerve transfer surgery targeting hand function without intraoperative or postoperative electrical stimulation. No additional patients will be enrolled in this group.
- Arm B: Standard nerve transfer surgery plus intraoperative and postoperative electrical stimulation: This is a prospectively enrolled group that will undergo standard nerve transfer surgery targeting hand function plus brief intraoperative electrical stimulation of the donor nerves and placement of a temporary peripheral nerve stimulator to allow postoperative electrical stimulation of the donor nerves for up to 60 days. All care provided, including the surgery, intraoperative electrical stimulation, postoperative electrical stimulation, and postoperative hand therapy, will be provided according to standard of care and is not considered experimental.
  Interventions: Device: Brief intraoperative electrical stimulation; Device: Temporary Postoperative Peripheral Nerve Stimulation

INTERVENTIONS:
Device: Brief intraoperative electrical stimulation — Intraoperative brief electrical stimulation (BES) will be performed using a handheld nerve stimulator (Checkpoint Guardian) to stimulate the donor nerves at 2 mA with a 200 µs pulse duration for 10 minutes per nerve.
  Other Names: Checkpoint Guardian Nerve Stimulator
  Groups: Arm B: Standard nerve transfer surgery plus intraoperative and postoperative electrical stimulation
Device: Temporary Postoperative Peripheral Nerve Stimulation — An implantable temporary peripheral nerve stimulator (SPRINT PNS System) will be placed during the surgery with one lead for each donor nerve. The implantable peripheral nerve stimulator will be programmed to optimize postoperative pain control on an individualized basis. The peripheral nerve stimulator will be explanted after 60 days, as is intended for this device.
  Other Names: SPRINT PNS System
  Groups: Arm B: Standard nerve transfer surgery plus intraoperative and postoperative electrical stimulation

SUMMARY:
The goal of this prospective observational study is to determine whether brief intraoperative electrical stimulation and temporary postoperative electrical stimulation improve motor and/or pain outcomes for patients with cervical spinal cord injury undergoing standard of care nerve transfer surgery to improve hand function.

The main hypotheses include:

Hypothesis #1: Brief intraoperative electrical stimulation of the donor nerves will result in improved motor outcomes (hand function) compared to standard nerve transfer surgery in patients with cervical spinal cord injuries.

Hypothesis #2: Placement of a temporary peripheral nerve stimulator for 60 days of postoperative electrical stimulation will result in improved pain outcomes compared to standard nerve transfer surgery in patients with cervical spinal cord injuries.

Researchers will prospectively enroll patients with cervical spinal cord injury and no hand function who will undergo standard of care nerve transfer surgery combined with standard of care brief intraoperative electrical stimulation and temporary postoperative electrical stimulation. Motor and pain outcomes will be compared to a retrospective group of patients who underwent nerve transfer surgery without intraoperative or postoperative electrical stimulation.

Participants will receive standard medical care (nothing experimental) as part of this study. Participants will:

* Have a preoperative assessment including physical examination, electrodiagnostic studies, functional electrical stimulation, and will complete questionnaires assessing function and quality of life
* Agree upon a surgical plan, including the specific nerve transfers to be performed and whether to include brief intraoperative electrical stimulation and/or temporary postoperative electrical stimulation before being considered for enrollment in the study
* Will undergo standard of care nerve transfer surgery, with at least one nerve transfer targeting improvement in hand function and will receive brief intraoperative electrical stimulation of the donor nerves and placement of a temporary peripheral nerve stimulator
* Will follow-up with the surgeon 3, 6, 12, 24, and 36 months after the surgery
* Will have a physical examination and will complete questionnaires at the postoperative visits
* Will participate in hand therapy following the operation
* Will be eligible for placement of a permanent peripheral nerve stimulator, depending on response to the temporary peripheral nerve stimulator.

DETAILED DESCRIPTION:
Background:

Spinal cord injury (SCI) is a major problem facing the general public, with particular relevance for military personnel, given the high frequency of SCI in combat-related injuries. Nerve transfer surgery is one option for restoring function in cervical SCI patients that shows great promise. A nerve transfer involves sacrificing a working nerve that arises from a spinal cord segment above the zone of injury and connecting it to a non-working nerve to reinnervate a target muscle. Restoring hand function is consistently rated by SCI patients, including our lived experience consultants, as most important, even more important than walking or bowel/bladder control. Nerve transfer surgery has been shown to be effective in restoring hand function, but additional improvements are needed, especially for restoring grasp. Furthermore, pain is a significant problem in patients with cervical SCI, with an unmet need for options for treating pain in these patients. Peripheral nerve electrical stimulation has been shown to improve axonal regeneration, muscle reinnervation, and motor recovery and has been used to treat neuropathic pain. Thus, the use of peripheral nerve electrical stimulation has the potential to simultaneously improve motor and pain outcomes in cervical SCI patients undergoing nerve transfer surgery but has never been studied.

Objectives/Hypotheses:

The investigators hypothesize that brief intraoperative electrical stimulation of the donor nerves will result in improved motor outcomes compared to standard nerve transfer. We also hypothesize that placement of a temporary peripheral nerve stimulator for 60 days of postoperative electrical stimulation will result in improved pain outcomes compared to standard nerve transfer.

Specific Aim:

Compare motor and pain outcomes for nerve transfers in cervical spinal cord injury patients with and without peripheral nerve stimulation.

Study Design:

A single center, unblinded, single arm, non-randomized, observational design will be utilized. A total of 10 patients with cervical spinal cord injury classified as ASIA A or B, with International Standards for Neurological Classification of Spinal Cord Injury neurological level of injury C6 or C7 will be recruited and will undergo standard end-to-end nerve transfer surgery targeting restoration of finger extension (posterior interosseous nerve recipient) and finger flexion (anterior interosseous nerve recipient) according to standard clinical care. The test intervention will consist of intraoperative brief electrical stimulation of the donor nerves and postoperative electrical stimulation via a temporary, implantable peripheral nerve stimulator. Intraoperative brief electrical stimulation (BES) will be performed using a handheld nerve stimulator to stimulate the donor nerves at 2 mA with a 200 µs pulse duration for 10 minutes. The implantable peripheral nerve stimulator will be programmed to optimize postoperative pain control on an individualized basis. The peripheral nerve stimulator will be explanted after 60 days, as is intended for this device. The primary outcomes will be manual motor testing graded on the Medical Research Council (MRC) scale (0-5) for the extensor digitorum communis (EDC) and flexor pollicis longus (FPL) and the Numeric Rating Scale (NRS) for pain in the treated extremity (0-10). Patients will have a baseline preoperative electrodiagnostic study and functional electrical stimulation performed, with the decision for surgery occurring as part of standard clinical care. Assessments will occur preoperatively and postoperatively at 3, 6, 12, 24, and 36 months. The researchers will compare these data to a retrospective group of patients who underwent similar nerve transfer surgery without intraoperative or postoperative electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical spinal cord injury, ASIA A or ASIA B
2. International Standards for Neurological Classification of Spinal Cord Injury neurological level of injury C6 or C7
3. Agreed upon surgical plan includes at least 1 nerve transfer targeting finger flexion with the anterior interosseous nerve as the recipient and at least 1 nerve transfer targeting finger extension with the posterior interosseous nerve as the recipient
4. Age 18-65 years
5. Mentally and physically able to comply with evaluations and assessments
6. Upper motor neuron pattern of injury in the recipient nerve with planned surgery 36 months or less from the time of injury OR lower motor neuron pattern of injury in the recipient nerve with planned surgery 9 months or less from the time of injury
7. Muscle grade at least 4+/5 on the Medical Research Council (MRC) scale in the territory of the donor nerve(s)
8. Stable function for at least 3 months (i.e., no ongoing recovery)
9. Non-operative rehabilitation for at least 3 months
10. Able to read and write in English at a level necessary to complete the questionnaires

Exclusion Criteria:

1. Contraindication to electrical stimulation, including any implanted electronic device such as a pacemaker or intrathecal drug delivery pump
2. Active infection at the operative site or systemic infection
3. Active malignancy
4. Pregnancy
5. Joint contractures or limited passive range of motion that would limit recovery of function
6. Lack of appropriate social support and/or infrastructure to commit to scheduled follow-up visits
7. Previous tendon transfer or other surgery for restoration of function following cervical spinal cord injury
8. Planned tendon transfer surgery or other surgery for restoration of function following cervical spinal cord injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical spinal cord injury patients aged 18-65 years with neurological level of injury C6 or C7 and limited or no hand function
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Composite Motor Score | 36 Months Postoperative
  A composite sum of the manual motor testing of the extensor digitorum communis and flexor pollicis longus muscles on the MRC scale (0-5 for each muscle, 0-10 composite score) will be calculated (composite motor score).
Percentage of Baseline Pain | 6 Months Postoperative
  The percentage of baseline pain in the operated limb will be calculated by dividing the postoperative NRS score by the baseline NRS score and multiplying by 100.

SECONDARY OUTCOMES:
Manual Motor Testing | 6, 12, and 24 Months Postoperative
  A composite sum of the manual motor testing of the extensor digitorum communis and flexor pollicis longus muscles on the MRC scale (0-5 for each muscle, 0-10 composite score) will be calculated (composite motor score).
Percentage of Baseline Pain | 3 Weeks, 12, 24, and 36 Months Postoperative
  The percentage of baseline pain in the operated limb will be calculated by dividing the postoperative NRS score by the baseline NRS score and multiplying by 100.
DASH Score | 6, 12, 24, and 36 Months Postoperative
  Patients will complete the Disabilities of the Arm, Shoulder, and Hand Questionnaire. The DASH score ranges from 0-100, with 0 representing normal function of the upper extremities and 100 representing maximal functional impairment.
MHQ Score | 6, 12, 24, and 36 Months Postoperative
  Patients will complete the Michigan Hand Questionnaire. The MHQ has a score range of 0-100, with 0 representing the worst hand function and 100 representing ideal hand function.
SCIM III Score | 6, 12, 24, and 36 Months Postoperative
  Patients will complete the Spinal Cord Independence Measure III Questionnaire. The SCIM III score ranges from 0-60, with 0 representing complete dependence and 60 representing complete independence.
Zung SDS | 6, 12, 24, and 36 Months Postoperative
  Patients will complete the Zung Self-rated Depression Scale Questionnaire. Zung SDS score ranges from 20-80, with normal (<50), mild depression (50 to 59), moderate to marked major depression (60 to 69), and severe to extreme major depression (>70).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Wilson, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University/Stanford Health Care, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No